CLINICAL TRIAL: NCT05347108
Title: Real-Time Accurate Pathology Inspection and Decompression Study: A Prospective Observational Study on the Correlation Between Duration of Pain and Changes in Pain Levels Following of a Laser Decompression Procedure to Relieve Spine Pain
Brief Title: Real-Time Accurate Pathology Inspection and Decompression Study
Acronym: RAPID
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: KM Clinical Research Group (Industry)
Responsible Party: Sponsor
Other Study IDs: CMC-01-2020
Record Dates: First submitted 2020-03-17; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Spine Injuries and Disorders; Pain, Chronic; Pain, Back; Pain, Neck; Radiculopathy
MeSH Terms: conditions — Disease; Chronic Pain; Back Pain; Neck Pain; Radiculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laser-assisted neural decompression (LAND) procedure — The LAND procedure is a minimally invasive spinal decompression procedure that uses a focused laser beam to reduce and remove disc herniations that are causing nerve compressions and impingements within the spinal canal. It is performed in an outpatient setting and the patient receives local anesthesia.
  The LAND procedure has been performed extensively over the past 2-years on hundreds of patients, so including patients that have previously had the surgery allows for additional data points and improved reporting.
  Other Names: LAND

SUMMARY:
The primary objective is changes in spine and lower limb pain following a laser-assisted neural decompression (LAND) procedure for the treatment of lumbar, thoracic, or cervical spine and/or extremity pain. Secondary objectives will be changes in quality of life, prescription pain medication use, and patient satisfaction with procedure outcomes.

DETAILED DESCRIPTION:
Objectives The primary objective is changes in spine and lower limb pain following a laser-assisted neural decompression (LAND) procedure for the treatment of lumbar, thoracic, or cervical spine and/or extremity pain. Secondary objectives will be changes in quality of life, prescription pain medication use, and patient satisfaction with procedure outcomes.

Design and Outcomes This is a prospective observational study to determine the degree to which a laser-assisted neural decompression (LAND) procedure relieves spine and extremity pain. Subjects will have elected to have the procedure are part of their standard of care in treating their spine and/or leg pain. Subjects will complete a baseline survey and two follow-up surveys at 3-months and 12-months after their procedure date.

Interventions and Duration There will be no study intervention. Subjects will only be monitored and evaluated for pre- and post-operative pain, quality of life, satisfaction, and medication use. Subjects will be followed for 12 months following their LAND procedure.

Sample Size and Population This study will last for 4 years starting February 10, 2020. There will be no maximum subject population size. We aim for a minimum population size of 1,500 in order to give statistical significance with results.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed spinal decompression procedure by their healthcare provider.
* Previous conservative care such as physical therapy or chiropractic care that failed to provide adequate pain relief.
* Willing and able to adhere to the protocol of the study including the survey timeline.
* Between the ages of 18-85 years.

Exclusion Criteria:

* Inability or unwillingness to give written informed consent.
* Not a candidate for the LAND procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of chronic spine and/or extremity pain that have tried at least 6 weeks of conservative care.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain assessed with visual analogue scale | 12-months
  Change in pain levels as measured by a visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- KMCRG, Lā‘ie, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No